CLINICAL TRIAL: NCT02522988
Title: The Use of an Open Label Placebo to Treat Cancer Related Fatigue in Cancer Survivors
Acronym: OLPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Theresa W. Hoenemeyer, Director, Education and Support Services, Comprehensive Cancer Center, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: X150506002
Record Dates: First submitted 2015-08-05; First posted 2015-08-14 (Estimated); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Fatigue
Keywords: cancer-related fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1a (Experimental): During the first 3-week period of the study, Group 1 will serve as the experimental arm and will receive the open-label placebo intervention. Group 1 participants will take 2 placebos in the morning and 2 placebos in the evening for 21 days.
  Interventions: Behavioral: Open-label placebo intervention
- Group 2a (No Intervention): During the first 3-week period of the study, Group 2 will serve as the comparator arm.
- Group 1b (No Intervention): During the last 3-week period of the study, Group 1 will serve as the comparator arm.
- Group 2b (Experimental): During the last 3-week period of the study, Group 2 will serve as the experimental arm and will receive the open-label placebo intervention.Group 2 participants will take 2 placebos in the morning and 2 placebos in the evening for 21 days.
  Interventions: Behavioral: Open-label placebo intervention

INTERVENTIONS:
Behavioral: Open-label placebo intervention — An open-label placebo intervention is an administered placebo that is fully disclosed to participants. It is delivered with a script that tells participants they are receiving placebos; placebos have been found to have effects that are comparable to some clinical treatments; placebos work because of conditioning, expectancies, interactions with care team and biochemical factors (i.e., dopamine, endorphins). Participants are given placebos to take for a 3-week period and will not receive placebos for a 4-week period (including a one-week washout period).
  Other Names: OLPI
  Arms: Group 1a; Group 2b

SUMMARY:
The purpose of this randomized-controlled, crossover pilot trial is to evaluate the feasibility, acceptability and effects of a non-deceptive (open-label) administration of placebo pills for treating cancer related fatigue (CRF). If significant effects are found, the investigators will later determine if the presence of a COMT Val18Met genotype variant predicts placebo responses.

DETAILED DESCRIPTION:
The investigators will conduct a pilot randomized-controlled, crossover trial to evaluate the feasibility, acceptability and effect of the open-label administration of placebo pills on CRF and associated psychosocial factors (e.g., emotional health, social health, quality of life, etc.) for cancer survivors (CSs) who have completed all cancer treatments yet continue to experience CRF. Additionally, in an exploratory manner, the investigators will collect DNA saliva specimens that will be analyzed for potential biomarkers that may predict placebo responses. To do this, investigators will use a 7-week, single site, two-parallel arm, randomized controlled crossover pilot study to determine the feasibility, acceptability and effects of an Open Label Placebo Intervention (OLPI) on CSs who completed cancer treatments at least 6 months prior to enrollment in the study and report a fatigue score of 4 or greater on a 0-10 scale. Investigators will enroll 80 eligible CS participants who will be randomized into two groups of 40 (Group1 and Group2 ). In this crossover study, participants in Group1, will receive an OLP (placebo pill) for 21-days (Period 1)and Group2 (Observational Controls) will not. After a 1-week washout period, Group2 will receive the OLP for 21-days (Period 2) and Group1 (Observational Controls) will not.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Stage II - IV cancer;
* Completed primary treatment 6months to 10 years;
* Report ≥4 (moderate fatigue) on a 0-10 fatigue severity rating scale;
* Agree not to change any medications or treatments during the study;
* Willingness to make 4 clinical site visits over the course of the 49-day study.

Exclusion Criteria:

* Stage 1 cancer;
* Uncontrolled diabetes;
* Uncontrolled COPD;
* Uncontrolled ischemic heart disease;
* Uncontrolled liver/kidney diseases;
* Uncontrolled autoimmune diseases;
* Uncontrolled psychiatric or cognitive diseases.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Enrollment Rate | End of Study (7 weeks)
  Unit of measure: number of enrollees / number of eligible participants as a measure of feasibility.
Accrual Rate as a Measure of Feasibility | End of Study (7 weeks)
  Unit of measure: number of accrued participants / recruitment goal (80); odds ration of expected time-to-first participant/ actual time-to-first patient enrollment.
Adherence Rate as a Measure of Feasibility | End of Study (7 weeks)
  Unit of measure: number of placebos taken / number prescribed (84)
Eligibility as a measure of Feasibility | End of Study (7 weeks)
  Unit of measure: number eligible for enrollment / number screened
Retention as a measure of Acceptability | End of Study (7 weeks)
  Unit of measure: number retained in study / number enrolled (goal = 75% of enrolled

SECONDARY OUTCOMES:
Measure of fatigue manifestation | Baseline, 3 weeks, 4 weeks and 7 weeks
  Units of measure: units on a scale using the Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF) instrument. 30-questions measure the global, somatic, affective, behavioral and cognitive manifestations of fatigue. Scale for items = 0 (not at all) - 4 (extremely)
Measurement of impact of fatigue on quality of life | Baseline, 3 weeks, 4 weeks and 7 weeks
  Unit of measure: units on a scale using the Medical Outcomes Study 36-Item Short Form (MOS-36) instrument. The 36-item instrument measures the impact of fatigue on vitality, physical functioning, emotional functioning, social functioning and mental health. Scale for items = 1 (limited a lot) - 3 (Not limited at all)
Measurement of the impact of fatigue on physical function | Baseline, 3 weeks, 4 weeks and 7 weeks
  Unit of measure: units on a scale using the FACT-Fatigue instrument; scale for impact is 0 = not at all; 10 = very much.
Measurement of fatigue severity | Baseline, 3 weeks, 4 weeks and 7 weeks
  Units of measure: units on a scale using the Fatigue Symptom Inventory (FSI) instrument. Scale = 0 (no fatigue / no interference) to 10 (extreme fatigue / interference)

OTHER OUTCOMES:
Test for the presence of a COMT Val158Met/Val or Val/Val variant gene | Baseline
  Investigators will collect and store saliva samples so, should significant OLPI effects be obtained, we can evaluate whether a potential biomarker (COMT Val158Met variant) associates with placebo responsiveness.

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Comprehensive Cancer Center, Birmingham, Alabama, United States

REFERENCES:
- [Background] Kelley JM, Kaptchuk TJ, Cusin C, Lipkin S, Fava M. Open-label placebo for major depressive disorder: a pilot randomized controlled trial. Psychother Psychosom. 2012;81(5):312-4. doi: 10.1159/000337053. Epub 2012 Aug 1. No abstract available. PMID 22854752
- [Background] Kam-Hansen S, Jakubowski M, Kelley JM, Kirsch I, Hoaglin DC, Kaptchuk TJ, Burstein R. Altered placebo and drug labeling changes the outcome of episodic migraine attacks. Sci Transl Med. 2014 Jan 8;6(218):218ra5. doi: 10.1126/scitranslmed.3006175. PMID 24401940
- [Result] Kaptchuk TJ, Friedlander E, Kelley JM, Sanchez MN, Kokkotou E, Singer JP, Kowalczykowski M, Miller FG, Kirsch I, Lembo AJ. Placebos without deception: a randomized controlled trial in irritable bowel syndrome. PLoS One. 2010 Dec 22;5(12):e15591. doi: 10.1371/journal.pone.0015591. PMID 21203519
- [Derived] Hoenemeyer TW, Baidwan NK, Hall K, Kaptchuk TJ, Fontaine KR, Mehta TS. An Exploratory Analysis of the Association Between Catechol-O-Methyltransferase and Response to a Randomized Open-Label Placebo Treatment for Cancer-Related Fatigue. Front Psychiatry. 2021 Jun 29;12:684556. doi: 10.3389/fpsyt.2021.684556. eCollection 2021. PMID 34267689
- See also: Open Label Placebo Effects — http://www.uab.edu/mix/stories/how-open-label-placebos-turn-fake-pills-into-real-treatment